CLINICAL TRIAL: NCT04799327
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled，Parallel-group Clinical Trial to Assess the Efficacy and Safety of Noiiglutide Injection in Obese Subjects Without Diabetes.
Brief Title: The Effect of SHR20004（Noiiglutide ） on Body Weight in Obese Subjects Without Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR20004-202
Record Dates: First submitted 2021-03-04; First posted 2021-03-16 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2021-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Parallel Assign to SHR20004 or placebo
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A (Experimental)
  Interventions: Drug: SHR20004
- Treatment group B (Experimental)
  Interventions: Drug: SHR20004
- Treatment group C (Experimental)
  Interventions: Drug: SHR20004
- Treatment group D (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SHR20004 — SHR20004：low dose
  Arms: Treatment group A
Drug: SHR20004 — SHR20004: medium dose
  Arms: Treatment group B
Drug: SHR20004 — SHR20004: high dose
  Arms: Treatment group C
Drug: placebo — Placebo
  Arms: Treatment group D

SUMMARY:
The study is being conducted to assess the efficacy and safety of SHR20004 on body weight in obese subjects without diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained prior to any trial-related activities
2. Body mass index (BMI) between 28 and 40 kg/m2(both inclusive)
3. Diet and exercise management for at least 3 months before screening and less than 5% change in body weight during the previous 3 months（self-reported）.

Exclusion Criteria:

1. History of endocrine disease or treatment that may significantly affect body weight prior to screening visit
2. History of diabetes
3. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 (MEN2)
4. History of pancreatitis
5. Previous surgical treatment of obesity
6. Screening calcitonin of 20 ng/L or above

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in body weight | Week 0, Week 24
  Change from baseline in body weight in kilograms

SECONDARY OUTCOMES:
Relative change from baseline in body weight(%) | Week 0, Week 24
  Relative change from baseline in body weight(%)
Proportion of subjects with body weight reduction greater than or equal to 5% and10% from baseline | Week 0, Week 24
  Proportion of subjects with body weight reduction greater than or equal to 5% and10% from baseline
Change from baseline in fasting plasma glucose | Week 0, Week 24
  Change from baseline in fasting plasma glucose in mmol/L
Change from baseline in fasting insulin | Week 0, Week 24
  Change from baseline in fasting insulin in μU/ml
Change from baseline in fasting C-peptide | Week 0, Week 24
  Change from baseline in fasting C-peptide in ng/ml
Change from baseline in fasting blood lipids | Week 0, Week 24
  Change from baseline in fasting blood lipids including TC\TG\H-DLC\L-DLC in mmol/L
Change from baseline in glycosylated hemoglobin | Week 0, Week 24
  Change from baseline in glycosylated hemoglobin(%)
Change from baseline in blood pressure | Week 0, Week 24
  Change from baseline in blood pressure in mmHg
Change from baseline in waist circumference | Week 0, Week 24
  Change from baseline in waist circumference in cm
Change from baseline in waist-to-hip ratio | Week 0, Week 24
  Change from baseline waist-to-hip ratio（waist and hip will be combined to report waist-to-hip ratio)
Change from baseline in BMI | Week 0, Week 24
  Change from baseline in BMI (weight and height will be combined to report BMI in kg/m^2)
Change from baseline in plasma glucose of 120 minutes after oral glucose tolerance test （OGTT） | Week 0, Week 24
  Change from baseline in plasma glucose of 120 minutes after OGTT in mmol/L
Change from baseline in insulin of 120 minutes after oral glucose tolerance test （OGTT） | Week 0, Week 24
  Change from baseline in insulin of 120 minutes after OGTT in μU/ml
Change from baseline in C-peptide of 120 minutes after oral glucose tolerance test （OGTT） | Week 0, Week 24
  Change from baseline in C-peptide of 120 minutes after OGTT in ng/ml
Change from baseline in AUC0-2h of plasma glucose during OGTT | Week 0, Week 24
  Change from baseline in AUC0-2h of plasma glucose during OGTT in mmol*hr/L
Change from baseline in AUC0-2h of insulin during OGTT | Week 0, Week 24
  Change from baseline in AUC0-2h of insulin during OGTT in μU*hr/ml
Change from baseline in AUC0-2h of C peptide during OGTT | Week 0, Week 24
  Change from baseline in AUC0-2h of C peptide during OGTT in ng*hr/ml
Percentage of subjects developing anti-drug antibody of SHR20004 | Week 0-25
Percentage of subjects with an Adverse events | Week 0-25
Percentage of subjects with Injection site reactions | Week 0-25
12-lead ECG | Week 0-25
  12-lead ECG in heart rate（beats）, PR interval（ms）, QT interval(ms), QTC interval(ms), and overall conclusion description
Concentration of SHR20004 in plasma at steady state | Week 8

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi